CLINICAL TRIAL: NCT05175768
Title: A Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Effect of Nicotinamide Mononucleotide (NMN) As an Adjuvant to Standard of Care (SOC) On Fatigue Associated With COVID-19 Infection
Brief Title: Study to Evaluate the Effect of Nicotinamide Mononucleotide (NMN) As an Adjuvant to Standard of Care (SOC) On Fatigue Associated With COVID-19 Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Required criteria of covid patient was not met
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: LGD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SE/210401/NM/COVID
Record Dates: First submitted 2021-12-28; First posted 2022-01-04 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Nicotinamide Mononucleotide; Leucine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotinamide Mononucleotide (Active Comparator): Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Interventions: Other: Nicotinamide Mononucleotide
- Nicotinamide Mononucleotide with L-Leucine (Active Comparator): Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Interventions: Other: Nicotinamide Mononucleotide with L-Leucine
- Placebo (Placebo Comparator): Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nicotinamide Mononucleotide — Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Arms: Nicotinamide Mononucleotide
Other: Nicotinamide Mononucleotide with L-Leucine — Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Arms: Nicotinamide Mononucleotide with L-Leucine
Other: Placebo — Two sachets to be taken orally after breakfast and Two sachets after lunch with water.
  Arms: Placebo

SUMMARY:
A Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Effect of Nicotinamide Mononucleotide (NMN) As an Adjuvant to Standard of Care (SOC) On Fatigue Associated with COVID-19 Infection

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥ 40 years of age at time of enrolment.
2. laboratory-confirmed diagnosis of SARS-CoV-2 infection as determined by RT-PCR/ Rapid antigen test/ any other test.
3. Hospitalized within 2 days from screening and exhibiting tachypnea with i) a respiratory rate (RR) > 30 breaths/min and ii) a SpO2 readings <90% on room air.
4. Less than or equal to 8 days from COVID-19 symptom onset prior to randomization. Symptoms are defined as one or more of the following: cough, fever, shortness of breath, chest pain, abdominal pain, nausea/vomiting, diarrhea, body aches, weakness/fatigue, chills/sweating, headache, confusion, sore throat, runny nose/congestion, loss of taste or smell, or any other COVID-19 symptoms as determined by the Investigator.
5. Requiring supplemental oxygen by i) mask or tongs, or ii) high-flow oxygen (WHO category 4 and 5).
6. Currently on the standard of care (SOC) for COVID-19 infection as prescribed by the investigator/ treating physician.
7. The SOC will include one or more of the following:

   * Anticoagulants
   * Antibiotics
   * Corticosteroid
   * Other treatment modalities (considered ethical by the investigator with the exception of protocol prohibited medications)
8. Patients previously diagnosed with hypertension or currently having a Systolic blood pressure ≥ 130mmHg and/or diastolic ≥ 85 mmHg
9. Abdominal obesity with a waist circumference > 88cm in women and > 102 cm in men.
10. Patients diagnosed with one or more conditions linked to metabolic syndrome, which includes:

    * Hyperlipidemia (as defined by a valid report of triglyceride level ≥ 150mg/dL or currently on medication for hyperlipidemia).
    * A valid report of HDL < 50mg/dL in women & < 40mg/dL in men.
    * Hyperglycemia (as defined by a valid report of Fasting glucose level ≥ 110 mg/dL or currently on anti-diabetic drugs)
11. Patients with an mBDS score ≥ 3.
12. Available for, and agrees to attend, all scheduled trial visits and assessments at the research site, and able to complete all assessments and documents contained in the research trial.
13. Naturally post-menopausal women with amenorrhea for 1 year will be eligible.
14. Females of childbearing potential should be either sexually inactive (abstinent) for 60 days prior to the first dose of the study, throughout the study and for 30 days after completion of the study, or be using one of the following acceptable methods of birth control:

    * Surgically sterile (bilateral tubal-ligation, hysterectomy, bilateral oophorectomy) for at least 90 days prior to the first dose of the study.
    * IUD in place for at least 60 days prior to the first dose of the study, throughout the study and for 30 days after completion of the study.
    * Hormonal contraceptives for at least 90 days prior to the first dose of the study, throughout the study, and for 30 days after study completion.

      * Changes to the method of birth control while participating in the study will be judged by the PI for acceptability.
15. Having given written informed consent by a legally acceptable representative to participate in the research trial.
16. Patients ready to abstain from Niacin and/or nicotinamide supplements.

Exclusion Criteria:

1. Hospitalized for more than 48 hours.
2. FBG levels ≥ 200 mg/dL
3. Known or suspected allergy to any of the ingredients in the investigational product or standardized meals.
4. Currently undergoing invasive mechanical ventilation (including venous ECMO) at the time of screening. (WHO category 6 and 7).
5. ALT/AST > 2.5 times the upper limit of normal or a history of decompensated cirrhosis.
6. Serum creatinine > 2 times the upper limit of normal.
7. Patients currently on monoclonal antibodies including antibody cocktails.
8. Patients for whom, in the opinion of the Investigator, progression to death is imminent and inevitable within the next 48 - 72 hours, irrespective of the provision of treatment.
9. Patients for whom, in the opinion of the Investigator, progression to mechanical ventilation is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment.
10. Possibility of the patient being discharged from hospital within 24 hours.
11. Participation in other anti-COVID-19 interventional trials.
12. Other known active infections or other clinical conditions (e.g., chronic obstructive pulmonary disease) that contraindicate aerosolized inhalation; coexisting pneumonia is allowed.
13. Patients with known instance of angina or myocardial infarction prior to 3 months of screening visit.
14. Patients with current or prior psychiatric illness, seizure disorders, autoimmune disorders, pre-existing severe cardiovascular disease and patients with prior transplants.
15. Females who are breast-feeding, lactating, pregnant or intending to become pregnant.
16. Diagnosed for hepatitis B, hepatitis C or uncontrolled HIV.
17. Presenting, in the opinion of the Investigator, a clinically significant abnormality with regard to the clinical examination and/or clinical chemistry screening parameters.
18. History of cancer in the last 5 years, or currently has cancer, as assessed by Investigator.
19. Has a history of, or current neurological (neurodegenerative diseases, epilepsy) or psychiatric pathology that may impact the participant's ability to comply with the requirements of the protocol, as assessed by Investigator.
20. Frequent consumption of alcohol (> 2 standard servings of alcohol/day on average).
21. History of (assessed by PI) or current tobacco use.
22. Patients with history of drug abuse (amphetamines, Cannabinoids, Cocaine and Opiates)
23. Inability to provide blood and/or urine samples.
24. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Multidimensional fatigue Inventory-20 | Upto 28 days
  Effect of on COVID-19 associated fatigue as assessed by the Multidimensional fatigue Inventory-20 scale.

SECONDARY OUTCOMES:
total number of days hospitalized | Upto 28 days
  Effect of IP on Duration of hospitalization by assessing the total number of days hospitalized.
Proportion of patients demonstrating clinical improvement | From baseline (day 0) to day of discharge (Upto 28 days)
  Effect of IP on the rate of recovery as assessed by the proportion of patients demonstrating clinical improvement defined by the WHO categories 0, 1, 2, or 3.
Modified Borg Dyspnoea Scale | Day 0, Day 4, Day of discharge, (Day 14 , Day 21) Optional, Day 28
  Effect of IP on breathlessness as assessed by the change in Modified Borg Dyspnoea Scale (mBDS) score
time taken to reach SPO2 ≥ 95% | Upto 28 days
  Effect of IP on time taken to reach SPO2 ≥ 95% without supplemental oxygen measured with pulse oximeter
the rate of recovered patients discharged | Upto 28 days
  Effect of IP on hospital discharge rate as assessed by the rate of recovered patients discharged from the hospital
rate of clinical deterioration | Upto 28 days
  Effect of IP on rate of clinical deterioration as assessed by the proportion of patients fulfilling WHO categories 6, 7 or 8
Viral load | Day 0, Day 4, Day of discharge (Upto 28 days)
  Effect of IP on SARS-CoV-2 viral load evaluated by RT-PCR (Ct Value)

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Dept of critical care medicine, new trauma centre, rajendra institute of medical sciences (RIMS),, Ranchi, Jharkhand
  - St. George's Hospital, Mumbai, Maharashtra
  - BAJ RR Hospital, Mumbai, Maharashtra
  - Pulse Multispeciality Hospital, Pune, Maharashtra
  - Jeevanrekha Multispeciality Hospital, Pune, Maharashtra
  - Ojas Multispeciality Hospital, Pune, Maharashtra
  - Krishna institute of medical sciences Deemed To Be University, Satara, Maharashtra
  - Acharya Vinoba Bhave Rural Hospital, Wardha, Maharashtra
  - Kalinga Institute of Medical Sciences (KIMS), Bhubaneswar, Odisha
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Jaipur National University Institute for Medical Science and Research Centre, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No